CLINICAL TRIAL: NCT06148584
Title: Feasibility and Acceptability of a Barbershop Based HIV Prevention Initiative Among Heterosexual Men in Kalangala Islands, Uganda: A Cluster Randomized Trial
Brief Title: Testing a Barbershop-based HIV Prevention Initiative Among Men
Acronym: TRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 111; UM1AI068619-17 (NIH)
Record Dates: First submitted 2023-10-27; First posted 2023-11-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: HIV; HIV Prevention; Barbershop; Uganda; Kalangala District; Heterosexual Men; HIV Education; HIV Self-test Kits; Peer Support; HIV Testing; HIV Risk Reduction Counseling; STI Testing
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Barbershops Group (Experimental): Participants recruited from intervention barbershops will receive the barbershop-based HIV prevention initiative. The trained barber will provide the following services during regular haircut services: general, status-neutral HIV education, HIV self-test kits, and information about where to receive HIV prevention services. The barber will also lead peer support group education every two months for clients enrolled in the study.
  Interventions: Behavioral: General, status-neutral HIV education; Diagnostic Test: HIV self-test kits; Other: Information about where to receive HIV prevention services; Behavioral: Barber-led peer support group education
- Control Barbershops Group (Active Comparator): Participants recruited from control barbershops will receive standard-of-care HIV prevention services which include facility-based HIV risk reduction counseling and testing and providing information about facility distributed HIV self-test kits.
  Interventions: Behavioral: Facility-based HIV risk reduction counseling; Diagnostic Test: Facility-based HIV testing; Other: Information about facility distributed HIV self-test kits; Diagnostic Test: STI testing

INTERVENTIONS:
Behavioral: General, status-neutral HIV education — General, status-neutral HIV education
  Arms: Intervention Barbershops Group
Diagnostic Test: HIV self-test kits — HIV self-test kits
  Arms: Intervention Barbershops Group
Other: Information about where to receive HIV prevention services — Information about where to receive HIV prevention services
  Arms: Intervention Barbershops Group
Behavioral: Barber-led peer support group education — Barber-led peer support group education
  Arms: Intervention Barbershops Group
Behavioral: Facility-based HIV risk reduction counseling — Facility-based HIV risk reduction counseling
  Arms: Control Barbershops Group
Diagnostic Test: Facility-based HIV testing — Facility-based HIV testing
  Arms: Control Barbershops Group
Other: Information about facility distributed HIV self-test kits — Information about facility distributed HIV self-test kits
  Arms: Control Barbershops Group
Diagnostic Test: STI testing — STI testing
  Arms: Control Barbershops Group

SUMMARY:
To test community-based approaches to engage heterosexual men at risk for HIV and specifically to assess the feasibility and acceptability of a barbershop based HIV prevention program.

DETAILED DESCRIPTION:
HPTN 111/TRIM is a cluster randomized study to assess the feasibility and acceptability of a barbershop-based HIV prevention program. Eighteen barbershops in Kalangala District, Uganda will be purposively selected to participate in the study and randomized 2:1 to provide the barbershop-based HIV prevention initiative (intervention) or the standard-of-care (control). Individual participants will be enrolled from the barbershops and receive intervention or control services based on their barbershop. The barbershop-based HIV prevention initiative will include barber provided status-neutral HIV education, HIV self-test kits, and information about where to receive HIV prevention services.

ELIGIBILITY:
Inclusion Criteria:

Persons who identify as a heterosexual male and meet all of the following criteria are eligible for inclusion in this study:

1. Age ≥ 16 years

   a. Any participants 16-17 years old will be enrolled following the Uganda National Council for Science and Technology (UNCST) guidelines for mature and emancipated minors
2. Able and willing to provide informed consent
3. Behaviorally vulnerable to HIV, based on self-report of at least one of the following in the last three months:

   1. Had condomless sex with a person of unknown HIV status or a person living with HIV
   2. Had more than one sexual partner
4. HIV negative per Ugandan Ministry of Health guidelines and the Study-specific Procedures (SSP) Manual
5. Is a regular customer at a participating barbershop as defined in the SSP Manual

Exclusion Criteria:

Persons who meet any of the following criteria will be excluded from this study:

1. Not planning to stay in the study catchment area in the next 12 months
2. Any other condition that in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Participants who report sex with other men will not be excluded from this study so long as they meet the inclusion and exclusion criteria listed above.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and acceptability of a barbershop based HIV prevention initiative | Week 26 and Week 52
  Consistent with this primary study objective, the following endpoint will be assessed from participants in the intervention group: Participant responses from surveys at Week 26 and Week 52 about acceptability of the intervention
To evaluate the feasibility and acceptability of a barbershop based HIV prevention initiative | Week 13, Week 26, Week 39, Week 52, Week 65
  Consistent with this primary study objective, the following endpoint will be assessed from participants in the intervention group: Barber responses from surveys about feasibility and acceptability of intervention
To evaluate the feasibility and acceptability of a barbershop based HIV prevention initiative | Week 26 and Week 52
  Consistent with this primary study objective, the following endpoint will be assessed from participants in the intervention group: Recruitment rates during enrollment and retention in study and barbershop activities at Week 26 and Week 52
To evaluate the feasibility and acceptability of a barbershop based HIV prevention initiative | Week 13, Week 26, Week 39, Week 52, Week 65
  Consistent with this primary study objective, the following endpoint will be assessed from participants in the intervention group: Frequency of barber-participant interactions
To evaluate the feasibility and acceptability of a barbershop based HIV prevention initiative | Week 13, Week 26, Week 39, Week 52, Week 65
  Consistent with this primary study objective, the following endpoint will be assessed from participants in the intervention group: Proportion of barber-participant interactions that include delivery of the intervention

SECONDARY OUTCOMES:
To compare completion of self-initiated HIV testing between intervention and control groups | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Self-report of HIV test conducted during the study follow-up
To evaluate the preliminary effectiveness of the intervention on change in risk behaviors associated with HIV acquisition | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Self-reported risk behaviors at Week 26 and Week 52, including condom use
To evaluate the preliminary effectiveness of the intervention on change in risk behaviors associated with HIV acquisition | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Self-reported risk behaviors at Week 26 and Week 52, including number of total sexual partners
To evaluate the preliminary effectiveness of the intervention on change in risk behaviors associated with HIV acquisition | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Self-reported risk behaviors at Week 26 and Week 52, including number of new sexual partners
To compare interest in or use of HIV prevention services between intervention and control groups | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Voluntary medical male circumcision (VMMC) during the study
To compare interest in or use of HIV prevention services between intervention and control groups | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Self-reported access to PEP care or use of PEP
To compare interest in or use of HIV prevention services between intervention and control groups | Week 26 and Week 52
  Consistent with this secondary study objective, the following endpoint will be assessed: Self-reported access to PrEP care or use of any PrEP method during the study
To assess the preliminary interest in Long-Acting PrEP (LAPrEP) among all participants | Week 52
  Consistent with this secondary study objective, the following endpoints will be assessed: Self-reported interest in LAPrEP at Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Lukyamuzi, MBChB, MPH, Study Chair — Makerere University, Johns Hopkins University Collaboration (MU-JHU); Brenda Gati Mirembe, MBChB, MscEpi, Study Chair — Makerere University, Johns Hopkins University Collaboration (MU-JHU)
Locations (1):
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT06148584/Prot_SAP_ICF_001.pdf